CLINICAL TRIAL: NCT01471899
Title: Randomized, Double Blind, Double Dummy To Non-Inferiority Comparison Of Ketorolac Tromethamine Oral Drops Versus Naproxen For Moderate to Severe Back Pain Treatment
Brief Title: Comparison Of Ketorolac Tromethamine Oral Drops Versus Naproxen For Moderate to Severe Back Pain Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTRGEMS0611
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Ketorolac Tromethamine; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naproxen (Active Comparator): 2 tablets every 8 hours for 4 days.
  Interventions: Drug: Naproxen
- Ketorolac Tromethamine (Experimental): 10 drops every 8 hours for 4 days
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — 10 drops each 8 hours for 4 days.
  Arms: Ketorolac Tromethamine
Drug: Naproxen — 2 tablets every 8 hours for 4 days
  Arms: Naproxen

SUMMARY:
The purpose of this study is to evaluate the non-inferiority clinical efficacy of two different drugs in the treatment of patients diagnosed with moderate to severe back pain treatment.

DETAILED DESCRIPTION:
* double-blind, double-dummy, non-inferiority, prospective, parallel group, intent to treat trial.
* Experiment duration: 04 days.
* 03 visits (days 0, 2 and 4).
* Efficacy will be evaluated for back pain relief based on visual analogic scale.
* Adverse events evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Consent of the patient or legal guardian.
* Men or women aged between 18 and 65.
* Diagnosis of acute low back pain with moderate to severe pain (Visual Analogic score greater than 4 cm)

Exclusion Criteria:

* fracture confirmed by X-ray
* Diagnosis of infection, fever,
* Pregnancy, lactation;
* Diagnosis of fibromyalgia;
* Hypersensitivity to ketorolac tromethamine, any of the ingredients of the formula or other Nonsteroidal anti-inflammatory

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment in back pain relief based on Visual Analogic Score (VAS). | 4 days
  The individual response rate to the relieve of pain is calculated by measuring VAS during the first and last visit.
  The response rate is calculated using the following formula:
  Response rate = (VASvi - VASvf) / VASvi
  Considering:
  * VASvi: VAS in the first visit;
  * VASvf: VAS at the last visit;

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences | day 4
  Adverse events will be collected and followed in order to evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Pérola Plaper, MD, Principal Investigator — Instituto do Coracao